CLINICAL TRIAL: NCT04177758
Title: A Prospective, Tripled-Blinded, Randomized Controlled Trial Evaluating Vitamin D3 Supplementation on Post-Operative Functional and Clinical Outcomes Following Total Knee Arthroplasty
Brief Title: Evaluating Vitamin D3 Supplement on Post-Op Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Denis Nam, M.D., M.Sc, Assistant Professor, Orthopedic Surgery, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19092704
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Results first posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Patients randomized to the control arm will receive placebo tablets and advised to consume their medication similar to the treatment arm.
  Interventions: Drug: Control
- Treatment (Experimental): Patients randomized to the experimental arm of the study will receive 50,000IU of vitamin D3 following surgery and asked to take the medication orally following surgery.
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Patients randomized to the experimental arm of the study will receive 50,000IU of vitamin D3 following surgery and asked to take the medication orally following surgery.
  Arms: Treatment
Drug: Control — Patients randomized to the control will receive a placebo
  Arms: Control

SUMMARY:
The aim of this study is to determine if vitamin D supplementation is associated with differences in short-term recovery in patients following total knee arthroplasty compared to patients who do not receive supplementation. If so, vitamin D supplementation has the potential to become widely incorporated into the routine care for patients undergoing knee replacements.

DETAILED DESCRIPTION:
Patients will be enrolled from the clinics of Dr. Denis Nam and Dr. Craig Della Valle, two fellowship-trained orthopedic surgeons in the division of Adult Reconstruction at Midwest Orthopedics at Rush University Medical Center. Study staff will screen the clinic schedule of each surgeon and will discuss the purposes of the investigation at the time of their visit. If the patient is willing to participate in the investigation, verbal and written consent will be obtained by the study staff. At the time of consenting, patients will also be asked to perform a TUG test and will be asked to complete the questions that comprise the functional component of the KSS score.

This study will be tripled-blinded, thus, the patients, clinicians, and research staff involved will be unaware of patient allocation during this study. Each patient will receive a study ID, and a computer randomization system will be used to allocate patients to receive either vitamin D3 or placebo based on their study ID. Only members of the Rush pharmacy staff will possess the list matching the study ID to the study group assignment, ensuring that the study remains triple-blinded and that study coordinators are unaware of a patient's assignment when he or she picks up the study medication from the pharmacy.

Patients randomized to the experimental arm of the study will receive 50,000IU of vitamin D3 following surgery and asked to take the medication orally following surgery. Vitamin D3 was selected over vitamin D2 as the former is less expensive and is more effective at raising serum 25-OH vitamin D levels than the latter. The regimen of 50,000IU given once was selected as this regimen has been previously used without side effects in previous studies and has been shown to be as effective as other regimens that utilize more frequent dosing with smaller doses. Patients randomized to the control arm will receive placebo tablets and advised to consume their medication similar to the treatment arm. Both groups of patients will receive their medications from the pharmacy at Rush Medical Center, which will be responsible for providing patients with the appropriate regimen. All patients will receive the same postoperative multimodal analgesic regimen that is normally administered to patients undergoing THA and TKA at Rush University Medical Center.

In accordance with current standard post-operative care, patients will be asked to follow-up with their surgeon in clinic at 3 weeks and 6 weeks following surgery. At these post-operative visits, patients will be asked to repeat the TUG test and the 17-questions of the functional component of the KSS score.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing primary total knee arthroplasty for osteoarthritis
* Age ≥ 18 years old
* Willingness to undergo randomization and return for all scheduled visits

Exclusion Criteria:

* Age > 80 years old
* American Society of Anesthesiologists (ASA) Score ≥ 4
* Other supplemental vitamin D or Calcium use including their analogs: ergocalciferol, calcitriol, dihydrotachysterol, and paricalcitol
* Current cancer
* Malabsorption syndromes
* Inability to take medications orally
* Renal impairment defined as a glomerular filtration rate (GFR) < 30 mL/minute or creatinine >1.3 mg/dL
* History of hypercalcemia defined as albumin-corrected hypercalcemia >12 mg/dL

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2022-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Nam, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Any patient undergoing primary total knee arthroplasty for osteoarthritis Age ≥ 18 years old Willingness to undergo randomization and return for all scheduled visits
Period: Overall Study
Arm/Group | Control | Treatment
Started | 69 | 68
Completed | 50 | 57
Not Completed | 19 | 11
Not completed — Lost to Follow-up | 19 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Treatment | Total
Number analyzed (Participants) | 50 | 57 | 107
Age, Categorical [Count of Participants; unit: Participants] — Population: Total patients allocated to treatment- (n=68), however, n=11 were removed, therefore, n=57 received allocated intervention
  Total patients allocated to placebo (control) (n=69). However, n=19 were removed, therefore, n=50 received allocated intervention.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 24 | 30 | 54
    >=65 years | 26 | 27 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.5 (8.5) | 63.7 (9.5) | 64.1 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 56
  Male | 23 | 28 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 57 | 107

OUTCOME MEASURES:

1. Primary Outcome: Knee Society Score (KSS), Functional Component (2012) at 3 Weeks Post Operative
Description: The functional component of the 2012 version of the knee society score at 3 weeks following surgery. Range 0-100. Assessed at 3 weeks following surgery, 3 weeks following surgery reported. For the 0-100 scale, Zero represents a worse outcome, deductions are taken away for using an assistive device and other physical exam factors. 100 would be the best score possible.
Time Frame: Assessed at 3 weeks following surgery
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 50 | 57
score on a scale | 46.94 [14 to 90] | 50.89 [5 to 100]

2. Primary Outcome: Knee Society Score (KSS) at 6 Weeks Following Surgery
Description: The functional component of the 2012 version of the knee society score at 6 weeks following surgery. Range 0-100. Assessed at 6 weeks following surgery, 6 weeks following surgery reported. For the 0-100 scale, Zero represents a worse outcome, deductions are taken away for using an assistive device and other physical exam factors. 100 would be the best score possible.
Time Frame: Assessed at 6 weeks following surgery reported
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Control | Treatment
Number analyzed (Participants) | 50 | 57
score on a scale | 55.43 [10.39 to 91] | 60.38 [22 to 100]

3. Secondary Outcome: Timed up and go Test at 3 Weeks Post Surgery
Description: A timed up and go (TUG) test at 3 weeks following surgery. The TUG test consists of measuring the time it takes for an individual to rise from a seated position in a chair, walk to a mark 3 meters away, turn around, come back, and sit in the same chair from which they started. Patients will be asked to perform the test twice at each of the aforementioned encounters. The use of any assistive devices such as cane or a walker) will also be noted.
Time Frame: Assessed at 3 weeks following surgery
Measure: Mean (Full Range); unit: seconds
Arm/Group | Control | Treatment
Number analyzed (Participants) | 50 | 57
seconds | 13.35 [7.42 to 31.94] | 13.46 [6.83 to 54.38]

4. Secondary Outcome: Timed up and go Test Difference From Baseline to 6 Weeks After Surgery
Description: A timed up and go (TUG) test difference from baseline and at 6 weeks following surgery. The TUG test consists of measuring the time it takes for an individual to rise from a seated position in a chair, walk to a mark 3 meters away, turn around, come back, and sit in the same chair from which they started. Patients will be asked to perform the test twice at each of the aforementioned encounters. The use of any assistive devices such as cane or a walker) will also be noted.
Time Frame: value at 6 weeks minus value at baseline
Measure: Mean (Full Range); unit: seconds
Arm/Group | Control | Treatment
Number analyzed (Participants) | 50 | 57
seconds | -0.9 [-14.5 to 11.7] | -0.3 [-14.2 to 9.3]

5. Secondary Outcome: Number of Participants With Complications
Description: Occurrence of any of the Knee Society's Standardized List of Complications
Time Frame: 6 weeks following surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Treatment
Number analyzed (Participants) | 50 | 57
Participants | 4 | 5

ADVERSE EVENTS:
Time Frame: Adverse events occurring 3 months post operative
Arm/Group | Control | Treatment
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/57
Other Adverse Events (participants affected / at risk) | 0/50 | 0/57

LIMITATIONS AND CAVEATS:
The dosing regimen included a one-time dose of 50,000IU vitamin D3, which may not be large enough to identify clinically significant differences. A higher than anticipated drop-out rate in this study occurred. Additionally, patients already taking vitamin D supplements were excluded from participation. We did not test patients for vitamin D deficiency preoperatively. We were unable to conduct a cost-analysis to support the cost-effectiveness of nonselective treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT04177758/Prot_SAP_000.pdf